CLINICAL TRIAL: NCT05704738
Title: A Phase 3, Randomized, 52-week, Placebo-controlled, Double-blind Study With Re-randomization to Assess the Efficacy, Safety, and Tolerability of Rocatinlimab (AMG 451) in Adolescent Subjects With Moderate-to-severe Atopic Dermatitis (AD) (ROCKET-ASTRO)
Brief Title: A Study to Evaluate Rocatinlimab (AMG 451) in Adolescent Participants With Moderate-to-severe Atopic Dermatitis (AD)
Acronym: ROCKET-ASTRO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20210145; 2022-501586-50 (Other: EUCTR)
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; AMG 451; KHK4083; Rocatinlimab
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Dose 1 (Experimental): Part 1 (Initial Period); Week 0 to Week 24: Rocatinlimab Dose 1 every 4 weeks (Q4W) for 24 weeks with loading dose at Week 2 (+ topical corticosteroids (TCS)/ topical calcineurin inhibitor (TCI) if within combination therapy cohort).
  Part 2 (Maintenance Period); Week 24 to Week 52: Part 1 Responders will be rerandomised at Week 24 to Rocatinlimab Dose 1 Q4W or every 8 weeks (Q8W) for 28 weeks (+ TCS/TCI if within combination therapy cohort).
  Interventions: Drug: Rocatinlimab
- Arm B: Dose 2 (Experimental): Part 1 (Initial Period); Week 0 to Week 24: Rocatinlimab Dose 2 Q4W for 24 weeks with loading dose at Week 2 (+TCS/TCI if within combination therapy cohort).
  Part 2 (Maintenance Period); Week 24 to Week 52: Part 1 Responders will be rerandomised at Week 24 to Rocatinlimab Dose 2 Q4W or Q8W for 28 weeks (with TCS/TCI if within combination therapy cohort).
  Interventions: Drug: Rocatinlimab
- Arm C: Placebo (Experimental): Part 1 (Initial Period); Week 0 to Week 24: Placebo Q4W for 24 weeks with loading dose at Week 2 (+TCS/TCI if within combination therapy cohort).
  Part 2 (Maintenance Period); Week 24 to Week 52: Part 1 Responders will be reassigned at Week 24 with Placebo Q4W for 28 weeks (with TCS/TCI if within combination therapy cohort).
  Interventions: Drug: Placebo
- Arm D: Open-Label Dose 1 (Experimental): Part 2; Week 24 to Week 52: Part 1 Non-Responders will be reassigned at Week 24 with Rocatinlimab Open-label Dose 1 Q4W for 28 weeks (with TCS/TCI if within combination therapy cohort). Participants in Arms A, B or C Maintenance Period will be reassigned with Rocatinlimab Open-label Dose 1 Q4W (with TCS/TCI if within combination therapy cohort) upon relapse after Week 24.
  Interventions: Drug: Rocatinlimab

INTERVENTIONS:
Drug: Rocatinlimab — Subcutaneous (SC) injection
  Other Names: AMG 451
  Arms: Arm A: Dose 1; Arm B: Dose 2; Arm D: Open-Label Dose 1
Drug: Placebo — SC injection
  Arms: Arm C: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of rocatinlimab in monotherapy and combination therapy treatment in adolescent participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 to < 18 years at Day 1.
* Diagnosis of AD (according to American Academy of Dermatology Consensus Criteria [Eichenfield et al, 2014]) that has been present for at least 12 months before signing of informed consent.
* Body weight ≥ 40 kg at screening.
* History of inadequate response to TCS of medium to higher potency (with or without TCI).
* EASI score ≥ 12 at initial screening.
* EASI score ≥ 16 at Day 1.
* vIGA-AD score ≥ 3.
* ≥10% body surface area of AD involvement.
* Worst pruritus NRS ≥ 4.

Exclusion Criteria:

* Treatment with a biological product within 12 weeks or 5 half-lives, whichever is longer, prior to Day 1.
* Treatment with any of the following medications or therapies within 4 weeks or 5 half-lives, whichever is longer, prior to Day 1:

  1. Systemic corticosteroids
  2. Non-biologic, non-targeted systemic immunosuppressants
  3. Phototherapy
  4. Oral or Topical Janus kinase inhibitors
* Treatment with any of the following medications or therapies within 1 week, prior to Day 1:

  1. TCS of any potency
  2. TCI
  3. Topical phosphodiesterase 4 inhibitors
  4. Other topical immunosuppressive agents

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 532 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Achievement of a Validated Investigator's Global Assessment for Atopic Dermatitis Score of 0 (Clear) or 1 (Almost Clear) with a ≥ 2 Point Reduction From Baseline (vIGA-AD 0/1) at Week 24 | Baseline and Week 24
Achievement of ≥ 75% Reduction From Baseline in EASI Score (EASI 75) at Week 24 | Baseline and Week 24

SECONDARY OUTCOMES:
Achievement of EASI 75 at Week 16 | Baseline and Week 16
Achievement of a vIGA-AD 0/1 at Week 16 | Baseline and Week 16
Achievement of a ≥ 4-point Reduction From Baseline in Weekly Average of Daily Worst Pruritus Numeric Rating Scale (NRS) Score at Week 16 in Participants with Baseline Weekly Average of Daily Worst Pruritus NRS Score ≥ 4 | Baseline and Week 16
Achievement of a ≥ 4-point Reduction From Baseline in Weekly Average of Daily Worst Pruritus NRS Score at Week 24 in Participants with Baseline Weekly Average of Daily Worst Pruritus NRS Score ≥ 4 | Baseline and Week 24
Achievement of ≥ 90% Reduction From Baseline in EASI Score (EASI 90) at Week 24 | Baseline and Week 24
Achievement of a ≥ 4-point Reduction From Baseline in Weekly Average of AD Skin Pain NRS Score at Week 24 in Participants with Baseline Weekly Average of AD Skin Pain NRS Score ≥ 4 | Baseline and Week 24
Achievement of a vIGA-AD Score of 1 with Presence of Only Barely Perceptible Erythema or vIGA-AD Score of 0 (revised Investigator's Global Assessment [rIGA™] 0/1) at Week 24 | Baseline and Week 24
Initiation of rescue therapy for AD at or before Week 16 | Baseline to Week 16
Initiation of rescue therapy for AD at or before Week 24 | Baseline to Week 24
Change From Baseline in Weekly Average of Daily Worst Pruritus NRS Score at Week 16 | Baseline to Week 16
Change From Baseline in Weekly Average of Daily Worst Pruritus NRS Score at Week 24 | Baseline to Week 24
Change From Baseline in Scoring of Atopic Dermatitis (SCORAD) Itch Visual Analog Scale (VAS) Score at Week 16 | Baseline to Week 16
Change From Baseline in SCORAD Itch VAS Score at Week 24 | Baseline to Week 24
Achievement of a ≥ 4-point Reduction from Baseline in Dermatology Life Quality Index (DLQI) Score at Week 24 in Participants with Baseline DLQI ≥ 4 in Participants ≥ 16 Years of Age at Enrollment | Baseline and Week 24
Change From Baseline in DLQI Score at Week 24 in Participants ≥ 16 Years of Age at Enrollment | Baseline to Week 24
Change From Baseline in CDLQI Score at Week 24 in Participants < 16 Years of Age at Enrollment | Baseline to Week 24
Achievement of a ≥ 4-point Reduction From Baseline in Patient Oriented Eczema Measure (POEM) Score at Week 24 in Participants with Baseline POEM Score ≥ 4 | Baseline and Week 24
Change From Baseline in POEM Score at Week 24 | Baseline to Week 24
Achievement of a ≥ 4-point Reduction From Baseline in Weekly Average of Daily AD Skin Pain NRS Score at Week 16 in Participants with Baseline Weekly Average of Daily AD Skin Pain NRS Score ≥ 4 | Baseline and Week 16
Change From Baseline in Weekly Average of Daily AD Skin Pain NRS Score at Week 24 | Baseline and Week 24
Change From Baseline in Weekly Average of Daily AD Skin Pain NRS Score at Week 16 | Baseline and Week 16
Achievement of a ≥ 3-point Reduction From Baseline in Weekly Average of Daily AD Skin Pain NRS Score at Week 24 in Participants with Baseline Weekly Average of Daily AD Skin Pain NRS Score ≥ 3 | Baseline and Week 24
Achievement of a ≥ 3-point Reduction From Baseline in Weekly Average of Daily AD Skin Pain NRS Score at Week 16 in Participants with Baseline Weekly Average of Daily AD Skin Pain NRS Score ≥ 3 | Baseline and Week 16
Change From Baseline in Weekly Average of Sleep Disturbance NRS Score at Week 24 | Baseline to Week 24
Achievement of a Hospital Anxiety and Depression Scale (HADS)-anxiety Subscale Score < 8 at Week 24 in Participants with Baseline HADS-anxiety Subscale Score ≥ 8 | Baseline and Week 24
Change From Baseline in HADS-anxiety Subscale Score at Week 24 | Baseline to Week 24
Achievement of a HADS-depression Subscale Score < 8 at Week 24 in Participants with Baseline HADS-depression Subscale Score ≥ 8 | Baseline and Week 24
Change From Baseline in HADS-depression Subscale Score at Week 24 | Baseline to Week 24
Achievement of a ≥ 8.7-point Reduction from Baseline in Severity SCORAD Score at Week 24 in Participants with Baseline SCORAD Score ≥ 8.7 | Baseline and Week 24

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (246):
- United States (98):
  - Cahaba Dermatology and Skin Health Center, Birmingham, Alabama
  - AllerVie Clinical Research- Cullman, Cullman, Alabama
  - Eclipse Clinical Research, Tucson, Arizona
  - Arkansas Research Trials, LLC, North Little Rock, Arkansas
  - Center for Dermatology Clinical Research Inc, Fremont, California
  - Doc1 Healthcare Systems Incorporated, Fullerton, California
  - Axon Clinical Research, Inglewood, California
  - Avance Clinical Trials, Laguna Niguel, California
  - Cura Clinical Research, Palmdale, California
  - Integrative Skin Science and Research, Sacramento, California
  - University of California at Davis Medical Center, Sacramento, California
  - Allergy and Asthma Medical Group and Research Center, San Diego, California
  - University of California at San Diego Rady Childrens Hospital San Diego, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Cura Clinical Research Sherman Oaks, Sherman Oaks, California
  - Velocity Clinical Research - Denver, Denver, Colorado
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Clinical Research of Brandon, Brandon, Florida
  - Academic Alliance in Dermatology - Saint Petersburg Office, Clearwater, Florida
  - Corazon United States of America, LLC doing business as Life Clinical Trials, Coral Springs, Florida
  - Palm Beach Dermatology Group, Delray Beach, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Glick Skin Institute, Margate, Florida
  - Miami Clinical Research, Miami, Florida
  - ara Professionals Limited Liability Corporation, Miami, Florida
  - Deluxe Health Care LLC, Miami Lakes, Florida
  - Savin Medical Group LLC, Miami Lakes, Florida
  - Angels Clinical Research Institute, Miami Lakes, Florida
  - Optimal Research Sites, LLC, Orange City, Florida
  - Clinical Associates of Orlando Limited Liability Company, Orlando, Florida
  - Clinical Research Investments, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Centricity Research Columbus, Columbus, Georgia
  - Advanced Medical Research PC, Sandy Springs, Georgia
  - Divine Dermatology and Aesthetics, Savannah, Georgia
  - McIntosh Clinic PC, Thomasville, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - NorthShore University HealthSystem Clinical Trials Center, Skokie, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Southern Indiana Clinical Trials, New Albany, Indiana
  - The Indiana Clinical Trials Center PC, Plainfield, Indiana
  - Equity Medical, Bowling Green, Kentucky
  - Kentucky Advanced Medical Research LLC, Murray, Kentucky
  - Industrial Medicine Associates Clinical Research Advanced Dermatology Care, Monroe, Louisiana
  - Aesthetic and Dermatology Center, Rockville, Maryland
  - Derm Associates, PC, Rockville, Maryland
  - Oakland Hills Dermatology, Auburn Hills, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Onyx Clinical Research, Flint, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Saint Louis University, St Louis, Missouri
  - Somnos Clinical Research, Lincoln, Nebraska
  - Skin Cancer and Dermatology Institute, Reno, Nevada
  - Allcutis Research, Portsmouth, New Hampshire
  - The Dermatology Center of New Jersey, Bridgewater, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Ace Clinical Trials, Brooklyn, New York
  - Empire Dermatology, East Syracuse, New York
  - Smart Medical Research Inc, Jackson Heights, New York
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Pioneer Clinical Research New York, New York, New York
  - Cornell University - Weill Cornell Medicine, New York, New York
  - Rochester Clinical Research, Rochester, New York
  - Yeshiva University - Montefiore Medical Center, The Bronx, New York
  - Duke South Durham, Durham, North Carolina
  - Optima Research, Boardman, Ohio
  - Apex Clinical Research Center LLC, Mayfield Heights, Ohio
  - Epic Medical Research - Oklahoma, Chickasha, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Dermatology and Aesthetics of Oklahoma, Oklahoma City, Oklahoma
  - Dermatology Research Center of Oklahoma, PLLC, Tulsa, Oklahoma
  - Essential Medical Research LLC, Tulsa, Oklahoma
  - Velocity Clinical Research - Grants Pass, Grants Pass, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Paddington Testing Company Inc, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Lifespan, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - National Allergy and Asthma Research, LLC, North Charleston, South Carolina
  - Coastal Pediatric Research, Summerville, South Carolina
  - HealthStar Physicians Dermatology, Morristown, Tennessee
  - The University of Texas Health Science Center at Houston, Bellaire, Texas
  - US Dermatology Partners Cedar Park, Cedar Park, Texas
  - Studies in Dermatology LLC, Cypress, Texas
  - MedCare Pharma - Houston, Houston, Texas
  - Tranquil Clinical Research, Houston, Texas
  - Sante Clinical Research, Kerrville, Texas
  - Long and Harris Dermatology, Lubbock, Texas
  - Sms Clinical Research Limited Liability Company, Mesquite, Texas
  - Sienna Dermatology Research, Missouri City, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Epiphany Dermatology, Southlake, Texas
  - Pioneer Research Solutions, Sugar Land, Texas
  - Tanner Clinic, Murray, Utah
  - Dermatology Research of Utah, dba Providence Dermatology, Providence, Utah
  - Jordan Valley Dermatology Center, South Jordan, Utah
  - Maria M Ona MD PC, Franklin, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
- Belgium (5):
  - Hopital Erasme, Brussels
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
  - Dermatologie Maldegem, Maldegem
- Brazil (11):
  - Centro do Diagnostico e Pesquisa da Osteoporose do Espirito Santo, Vitória, Espírito Santo
  - Clinica Instituto Bahiano de Imunoterapia - Medicina, Reumatologia e Dermatologia ltda, Salvador, Estado de Bahia
  - Centro de Pesquisa Clínica da Universidade de Belo Horizonte - Unibh, Belo Horizonte, Minas Gerais
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Cecip Centro Est Clin Int Paulista, Jaú, São Paulo
  - Le Plume Dermatologia- Clinica de Dermatologia Dra Beatriz Elias Eirelli, Ribeirão Preto, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Instituto Pesquisa e Ensino em Saúde Infantil, São Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
  - IBPClin Instituto Brasil de Pesquisa Clinica, Rio de Janeiro
- Canada (6):
  - Rejuvenation Dermatology Laser Calgary North, Calgary, Alberta
  - Lynderm Research Inc, Markham, Ontario
  - Dr SK Siddha Medicine Professional Corporation, Newmarket, Ontario
  - Allergy Research Canada Incorporated, Niagara Falls, Ontario
  - XLR8 Medical Research, Incorporated, Windsor, Ontario
  - Skinsense Medical Research, Saskatoon, Saskatchewan
- Chile (5):
  - Centro Dermatologico Dermisur, Osorno
  - Centro Medico Skinmed Spa, Santiago
  - Clinica Dermacross SA, Santiago
  - Fundacion Innovacion Cardiovascular, Santiago
  - Centro Internacional de Estudios Clinicos, Santiago
- China (24):
  - Childrens Hospital Capital Institute of Pediatrics, Beijing, Beijing Municipality
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - Beijing Childrens Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Childrens Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital Sun-Yat Sen University, Guangzhou, Guangdong
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - Nanyang First Peoples Hospital, Nanyang, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangyin Hospital of Traditional Chinese Medicine, Jiangyin, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Dalian Women and Childrens Medical Group, Dalian, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - Chengdu Second Peoples Hospital, Chengdu, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Kunming Childrens Hospital, Kunming, Yunnan
  - Affiliated Hangzhou First Peoples Hospital School of Medicine Westlake University, Hangzhou, Zhejiang
  - Ningbo NO 2 Hospital, Ningbo, Zhejiang
  - Taizhou Central Hospital, Taizhou, Zhejiang
  - Hunan Childrens Hospital, Changsha
  - Shenzhen Childrens Hospital, Shenzhen
- Croatia (5):
  - Special Hospital for Medical Rehabilitation Naftalan, Ivanić-Grad
  - University Hospital Centre Osijek, Osijek
  - Children s Hospital Zagreb, Zagreb
  - Sestre milosrdnice University Hospital Center, Zagreb
  - University Hospital Centre Zagreb, Zagreb
- France (7):
  - Hopital Prive d Antony, Antony
  - Centre Hospitalier Regional Universitaire Brest Hopital Morvan, Brest
  - Hôpital Saint-Joseph, Marseille
  - Centre Hospitalier Universitaire de Nantes Hôtel Dieu, Nantes
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - Centre Hospitalier Universitaire de Rouen - Hôpital Charles Nicolle, Rouen
  - Centre Hospitalier Universitaire de Toulouse, Hopital Larrey, Toulouse
- Germany (8):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Universitaetsklinikum Bonn, Bonn
  - Rosenpark Research GmbH, Darmstadt
  - Universitaetsklinikum Dresden, Dresden
  - Universitaetsklinikum Erlangen, Erlangen
  - Klinikum und Fachbereich Medizin Johann Wolfgang Goethe-Universitaet Frankfurt am Main, Frankfurt am Main
  - Velocity Clinical Research, Leipzig
  - Johannes Gutenberg Universitaet Mainz, Mainz
- Greece (4):
  - Athens Naval Hospital, Athens
  - Athens General Childrens Hospital Panagioti And Aglaia Kyriakou, Athens
  - Thoracic General Hospital Of Athens Sotiria, Athens
  - Ippokratio General Hospital of Thessaloniki, Thessaloniki
- Hungary (4):
  - Clinexpert Kft, Budapest
  - Derma-B Egeszsegugyi es Szolgaltato Kft, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár
- Israel (3):
  - Soroka Medical Center, Bear Sheva
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Italy (4):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli, Napoli
  - Azienda Ospedaliera di Perugia Ospedale Santa Maria della Misericordia, Perugia
  - Presidio Molinette Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Torino
- Japan (16):
  - Central Clinic, Nagoya, Aichi-ken
  - Miyata Dermatology Clinic, Matsudo-shi, Chiba
  - Matsuo Clinic, Fukuoka, Fukuoka
  - Asahikawa City Hospital, Asahikawa-shi, Hokkaido
  - Takagi Dermatological Clinic, Obihiro-shi, Hokkaido
  - Yoshimura Child Clinic, Akashi-shi, Hyōgo
  - Katahira Dermatology Urology Clinic, Kagoshima, Kagoshima-ken
  - Nomura Dermatology Clinic, Yokohama, Kanagawa
  - Yokohama City Minato Red Cross Hospital, Yokohama, Kanagawa
  - Jouzan Hihuka Hinyoukika Clinic, Kumamoto, Kumamoto
  - Suizenji Dermatology Clinic, Kumamoto, Kumamoto
  - Yoshioka Dermatology Clinic, Neyagawa, Osaka
  - Dermatology and Ophthalmology Kume Clinic, Sakai-shi, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Naoko Dermatology Clinic, Setagaya-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
- Phylasis Clinicas Research Toluca, Toluca, Mexico
- Poland (16):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - AKK Medical Spolka z ograniczona odpowiedzialnoscia Centrum Medyczne Tu sie leczy, Gdansk
  - GynCentrum Sp zoo NZOZ Holsamed, Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - Specjalistyczny Gabinet Dermatologiczny Aplikacyjno-Badawczy Marek Brzewski Pawel Brzewski SpCywilna, Krakow
  - Diamond Clinic Spolka z Ograniczona Odpowiedzialnoscia Diamond Medical Center, Krakow
  - AppleTreeClinics Network Spzoo, Lodz
  - Amicare Spolka z ograniczona odpowiedzialnoscia Spolka Komandytowa Amicare Centrum Medyczne, Lodz
  - Clinical Best Solutions Sp zoo Spolka Komandytowa, Lublin
  - Centrum Zdrowia Dziecka i Rodziny Im Jana Pawla II w Sosnowcu Osrodek Badan Klinicznych, Sosnowiec
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Spzoo, Tarnów
  - Klinika Osipowicz and Turkowski Sp zoo, Warsaw
  - High Med Przychodnia Specjalistyczna, Warsaw
  - Klinika Ambroziak Dermatologia, Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
  - Dermatologiczna Praktyka Lekarska Michal Torz Dermaceum Centrum Badan Klinicznych, Wroclaw
- Puerto Rico (2):
  - Clinical Research of Puerto Rico, San Juan
  - Gcm Medical Group, Psc, San Juan
- Romania (3):
  - Dr Leventer Centre Clinica Dermatologie Bucuresti, Bucharest
  - Derma Cluj, Cluj-Napoca
  - Institutul Regional de Gastroenterologie si Hepatologie Prof Dr Octavian Fodor, Cluj-Napoca
- South Korea (11):
  - Korea University Ansan Hospital, Ansansi, Gyeonggido
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - National Medical Center, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (5):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Catalonia
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario La Paz, Madrid
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Thailand (4):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Thammasat University Hospital, Pathum Thani

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Guttman-Yassky E, Simpson E, Bissonnette R, Eichenfield LF, Kabashima K, Luna PC, Hercogova JT, Spelman L, Worm M, Esfandiari E, Arai T, Mano H, Charuworn P, Wang A, Kricorian G. ROCKET: a phase 3 program evaluating the efficacy and safety of rocatinlimab in moderate-to-severe atopic dermatitis. Immunotherapy. 2025 Feb;17(2):83-94. doi: 10.1080/1750743X.2025.2464528. Epub 2025 Feb 26. PMID 40012373
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com